CLINICAL TRIAL: NCT02061956
Title: A Simple Prognostic Scoring System for Patients Receiving Transarterial Chemoembolization for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Professor, Sun Yat-sen University
Other Study IDs: HCC-0014
Record Dates: First submitted 2014-01-22; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HCC received TACE: Patients with HCC in cancer center, Sun Yat-sen University received TACE between 2011.01-2011.12

SUMMARY:
Hepatocellular carcinoma (HCC) is the 6th most common cancer worldwide and the third most frequent cause of death of cancer.Although with the development of medical science, more and more patients diagnose HCC at early stage, a lot of patients with HCC still continue to present with multiple tumors or port vein thrombosis. According to AASLD guidelines, these patients could received transcatheter arterial chemoembolization (TACE) or new agents as initial treatment. However, the intermediate group comprises a wide spectrum in terms of liver function and extent of tumour, and this may explain the large differences in survival reported for individual series.

A simple, pragmatic and reliable prognostic index based on objective measures would be of value in providing information to patients, for stratifying patients entering clinical trials and in making meaningful comparisons between series reported in the literature.The aims of our study were (i) to identify predictors of survival in a cohort of patients undergoing TACE or TAE for unresectable HCC, (ii) to develop and validate a simple scoring system and (iii) to compare the new scoring system with the most frequently used prognostic systems for its ability to separate high- and low-risk patients.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the 6th most common cancer worldwide and the third most frequent cause of death of cancer. The 2005 guidelines of the American Association for the Study of Liver Diseases (AASLD) for HCC states that hepatic resection(HR) can be offered to patients with a solitary lesion if they are non-cirrhotic, or have cirrhosis but still have well-preserved liver function. With the improvement of surgical technique and perioperative care, the surgical mortality for HCC resection can be reduced to less than 1%, and the 5-year overall survival can exceed 50%. Although with the development of medical science, more and more patients diagnose HCC at early stage, a lot of patients with HCC still continue to present with multiple tumors or port vein thrombosis. According to AASLD guidelines, these patients could received transcatheter arterial chemoembolization (TACE) or new agents as initial treatment. However, the intermediate group comprises a wide spectrum in terms of liver function and extent of tumour, and this may explain the large differences in survival reported for individual series.

A simple, pragmatic and reliable prognostic index based on objective measures would be of value in providing information to patients, for stratifying patients entering clinical trials and in making meaningful comparisons between series reported in the literature.The aims of our study were (i) to identify predictors of survival in a cohort of patients undergoing TACE or TAE for unresectable HCC, (ii) to develop and validate a simple scoring system and (iii) to compare the new scoring system with the most frequently used prognostic systems for its ability to separate high- and low-risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18-75 years;
2. Child-Pugh A or B liver function;
3. Eastern Cooperative Oncology Group (ECOG) performance scores ≤2;
4. HCC with no previous treatment;

Exclusion Criteria:

1. severe coagulopathy (prothrombin activity <40% or a platelet count of <40,000/mm3);
2. Child-Pugh C liver function or evidence of hepatic decompensation including ascites, esophageal or gastric variceal bleeding, or hepatic encephalopathy;

(4) ECOG scores 3-4 (5) combined with serious diseases of other organs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable HCC received TACE.The diagnosis of HCC was confirmed by either histology, cytology, elevated alpha-fetoprotein (AFP, >400 ng/mL), or by typical radiological appearance.
Sampling Method: Probability Sample
Enrollment: 647 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | 1 year
  1-year overall survival

SECONDARY OUTCOMES:
Safety | 1 month
  1 month mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China